CLINICAL TRIAL: NCT02091648
Title: A Pilot Stress Management Intervention for High Risk Children With Asthma
Brief Title: A Pilot Stress Management Intervention Study for High Risk Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Anna L. Marsland, Associate Professor of Psychology and Nursing, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34HL107613 (NIH)
Record Dates: First submitted 2014-03-04; First posted 2014-03-19 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Asthma
Keywords: Asthma; Stress; Children; Psychosocial Factors; Relaxation; Stress management
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I Can Cope Intervention (Experimental): Participants randomized to the "I Can Cope" condition will receive 6 face-to-face individualized sessions over a 2-month period. Each session will last 50 minutes and take place at the child's school either during approved times during the school day or as part of the after-school program. Sessions are psychoeducational and experiential and include opportunities for the child with asthma to: (1) learn about the pathophysiology of asthma; (2) understand the biological impact of stress on the body; (3) learn the relationship among thoughts, feelings, actions, and asthma; (4) acquire a set of coping skills to help deal with asthma-related and day-to-day stressors in their lives, and (5) receive training in biofeedback-assisted relaxation techniques.
  Interventions: Behavioral: I Can Cope Intervention
- Standard Education Intervention (Active Comparator): this group will receive the standard American Lung Association "Open Airways for Schools" program. This program includes six 40-minute sessions covering the National Heart Lung and Blood Institute recommendations for asthma education.
  Interventions: Behavioral: Standard Education Intervention
- No treatment control (No Intervention): This group will receive no treatment during the course of the study and will have the option to receive the "Open Airways" program after their participation in the study is complete.

INTERVENTIONS:
Behavioral: I Can Cope Intervention — Participants randomized to the "I Can Cope" condition will receive 6 face-to-face individualized sessions over a 2-month period. Each session will last 50 minutes and take place at the child's school either during approved times during the school day or as part of the after-school program. Sessions are psychoeducational and experiential and include opportunities for the child with asthma to: (1) learn about the pathophysiology of asthma; (2) understand the biological impact of stress on the body; (3) learn the relationship among thoughts, feelings, actions, and asthma; (4) acquire a set of coping skills to help deal with asthma-related and day-to-day stressors in their lives, and (5) receive training in biofeedback-assisted relaxation techniques.
  Arms: I Can Cope Intervention
Behavioral: Standard Education Intervention — This group will receive the standard American Lung Association (ALA)"Open Airways for Schools" program. This program includes six 40-minute sessions covering the National Heart Lung and Blood Institute's recommendations for asthma education.
  Other Names: Open Airways for Schools Program
  Arms: Standard Education Intervention

SUMMARY:
The purpose of the proposed study is to conduct a randomized controlled pilot trial of a school-based stress management and coping skills training program among a sample of economically disadvantaged urban 8- to 12-year-old school children with physician-confirmed asthma. The investigators aim (1) to establish feasibility of this approach by recruiting from different schools and (2) to learn whether individuals assigned to receive the intervention show improvements in psychological function, decreases in lung inflammation, and related improvements in asthma health when compared with disease severity-matched peers who receive education-only or standard care.

ELIGIBILITY:
Inclusion Criteria:

* In grades 3 through 8 and attending one of the 11 participating public schools
* Age 8 through 14 years
* Qualify for the free or reduced cost school lunch program in Pennsylvania (families that receive food stamps or have an annual income of < $40,900).
* Meets National Heart Lung and Blood Institute (NHLBI, 2007) criteria for any asthma diagnosis EXCEPT mild, intermittent asthma, as confirmed by the study physician using NHLBI Guidelines for the Diagnosis and Management of Asthma (http://www.nhlbi.nih.gov/guidelines/asthma/asthsumm.pdf, page 40).
* Has a parent or legal guardian who is willing to participate in the study
* Fluent in English (i.e., have commonly used English in everyday speaking and reading for at least 10 years)

Exclusion Criteria:

* History of a chronic illness in addition to asthma (determined by parent or guardian report)
* Prescribed medications other than for asthma
* Mental retardation or significant developmental delay
* Inability to speak or understand English
* A diagnosis of mild, intermittent asthma as determined using NHLBI (2007) criteria (see above)
* Age less then 8 years or greater than 14 years
* Not in grades 3 through 8
* Not qualifying for free or reduced cost school lunches in Pennsylvania
* No parent or legal guardian who is willing to participate

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Proportion of Eligible Children who Participate in Study | End of enrollment: estimated 2 years after beginning active enrollment.
  A measure of the feasibility of offering the "I Can Cope" intervention trial to socioeconomically disadvantaged 8-14 year-old children with physician-confirmed asthma in urban schools.
Participant Drop-out Rates | After final outcome measures are collected: up to 2 1/2 years from beginning of active enrollment.
  A measure of the feasibility of offering the "I Can Cope" intervention trial to socioeconomically disadvantaged 8-14 year-old children with physician-confirmed asthma in urban schools.
Session Completion Rates | After final participant has completed study: estimated 2 1/2 years after beginning active enrollement.
  A measure of the feasibility of offering the "I Can Cope" intervention trial to socioeconomically disadvantaged 8-14 year-old children with physician-confirmed asthma in urban schools.
Program Satisfaction Survey | End of Study Participation: up to 5 months from initial enrollment.
Barriers to offering the Intervention in Selected Schools | End of enrollment: estimated 2 years after beginning active enrollment.
Child Depression Inventory | Pre and Post Intervention: baseline, up to 4 months later.
  Assess change in symptoms of depression.
State-Trait Anxiety Inventory for Children | Pre and Post Intervention: baseline, up to 4 months later.
  Assess change in symptoms of anxiety and depression.
Perceived Stress Scale | Pre and post intervention: baseline, up to 4 months later.
  Assess change in the degree to which the child perceives current demands as stressful and exceeding his or her ability to cope.
Pediatric Asthma Quality of Life Questionnaire | Pre and Post Intervention: baseline, up to 4 months later.
  Assesses asthma-related quality of life.
Asthma Self-Management Scale | Pre and Post Intervention: baseline, up to 4 months later.
  Parent and child participants will complete the which assesses beliefs that they can perform behaviors to alleviate the child's asthma, including behaviors associated with symptom prevention (e.g., getting to doctor, using medication, and avoiding allergens) as well as symptom management (e.g., staying calm, controlling symptoms, deciding how to manage symptoms).
KIDCOPE | Pre and Post Intervention: baseline, up to 4 months later.
  Child participants will complete the Kidcope a 10-item measure of different coping strategies.
Measure of Current Status (MOCS - Adapted) | Pre and Post Intervention: baseline, up to 4 months later.
  In order to measure the effectiveness of stress management training, child participants will complete an adapted version of the 10-item Measure of Current Status assessing perceived self-efficacy for skills targeted by the intervention: the ability to relax, to recognize stress-inducing situations, to be assertive about needs, and to choose appropriate coping responses.
Change in Asthma Health from Baseline | Pre to post-intervention: baseline, up to 4 months later.
  The magnitude of intervention-related improvements in the child's asthma health will be measured by change in pulmonary function, exhaled levels of nitric oxide, and symptoms of asthma, as well as number of medical visits, and school absenteeism.

SECONDARY OUTCOMES:
Life Events Questionnaire | Baseline
  Assesses life events that have had a negative impact on the child's psychological state.

CONTACTS AND LOCATIONS:
Overall Officials: Anna L. Marsland, Ph.D., R.N., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Long KA, Ewing LJ, Cohen S, Skoner D, Gentile D, Koehrsen J, Howe C, Thompson AL, Rosen RK, Ganley M, Marsland AL. Preliminary evidence for the feasibility of a stress management intervention for 7- to 12-year-olds with asthma. J Asthma. 2011 Mar;48(2):162-70. doi: 10.3109/02770903.2011.554941. PMID 21332379
- [Derived] Marsland AL, Gentile D, Hinze-Crout A, von Stauffenberg C, Rosen RK, Tavares A, Votruba-Drzal E, Cohen S, McQuaid EL, Ewing LJ. A randomized pilot trial of a school-based psychoeducational intervention for children with asthma. Clin Exp Allergy. 2019 May;49(5):591-602. doi: 10.1111/cea.13337. Epub 2019 Feb 8. PMID 30657230